CLINICAL TRIAL: NCT03512808
Title: A Single-dose, Comparative Bioavailability Study of Two Formulations of Ursodiol 500mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-4052
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Healthy
MeSH Terms: interventions — Ursodeoxycholic Acid; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ursodiol 500mg tablets (Experimental): Ursodiol 500mg tablets followed by Urso Forte 500mg tablets
  Interventions: Drug: Ursodiol 500 MG
- Urso Forte 500mg tablets (Active Comparator): Urso forte 500mg tablets followed by Ursodiol 500mg tablets
  Interventions: Drug: Urso Forte 500Mg Tablet

INTERVENTIONS:
Drug: Ursodiol 500 MG — Ursodiol 500mg tablets followed by Urso Forte 500mg tablets
  Arms: Ursodiol 500mg tablets
Drug: Urso Forte 500Mg Tablet — Urso forte 500mg tablets followed by Ursodiol 500mg tablets
  Arms: Urso Forte 500mg tablets

SUMMARY:
A single-dose, comparative bioavailability study of two formulations of ursodiol 500mg tablets under fasting conditions

DETAILED DESCRIPTION:
A single-dose, comparative bioavailability study of two formulations of ursodiol 500mg tablets under fasting conditions: open label, single-dose, randomized, two-period, two-treatment, two-sequence, crossover, comparative bioavailability study

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects, 18 years of age or older
* BMI ≥ 19.0 and ≤ 30.0 kg/m2.
* Females who participate in this study will be of chilbearing or non-childbearing potential

Exclusion Criteria:

• Know history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the investigator, would jeopardized the safety of the subject or impact the validity of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0-72 hours
Area under the plasma concentration versus time curve (AUC) | 0-72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Pharma medica research Inc., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No